CLINICAL TRIAL: NCT05712148
Title: Suprachoroidal Spheroidal Mesenchymal Stem Cell Implantation in Retinitis Pigmentosa: Clinical Results of 6 Months Follow-up
Brief Title: Spheroidal Mesenchymal Stem Cells in Retinitis Pigmentosa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Berna Özkan, Professor, Acibadem University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 56733164/203 E.3858
Record Dates: First submitted 2023-01-16; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Retinitis Pigmentosa; Stem Cell Transplant
Keywords: Retinitis pigmentosa; Mesenchymal stem cells; Spheroids; Suprachoroidal implantation
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Retinitis Pigmentosa patients (Experimental): Suprachoroidal mesenchymal stem cell implanted Retinitis pigmentosa patients
  Interventions: Biological: Stem cell implantation

INTERVENTIONS:
Biological: Stem cell implantation — Suprachoridal mesenchymal spheroidal stem cell implantation

SUMMARY:
Purpose: This prospective clinical case series aimed to evaluate the effect of suprachoroidal implantation of mesenchymal stem cells (MSCs) in the form of spheroids as a stem cell therapy for retinitis pigmentosa (RP) patients with relatively good visual acuity.

Methods: Fifteen eyes of 15 patients with RP who received suprachoroidal implantation of MSCs in the form of spheroids were included. Best corrected visual acuity (BCVA), 10-2 and 30-2 visual field examination and multifocal electroretinography (mfERG) recordings were recorded at baseline, postoperative first, third- and sixth-months during follow-up.

DETAILED DESCRIPTION:
A prospective clinical trial was conducted in patients with RP at the department of ophthalmology, Acibadem University, Medical school. The study was approved by the Review Board of Cell, Organ and Tissue Transplantation Department of Turkish Ministry of Health. The study was performed in accordance with the Declaration of Helsinki.

Patient Evaluation Fifteen patients with clinical and genetic diagnoses of RP were included in the study. Patients underwent ophthalmic examination including best corrected visual acuity (BCVA), intraocular pressure, anterior segment examination and dilated fundus examination (with topical tropicamide %1 and phenylephrine 2.5%). Each eye underwent spectral domain OCT scanning with Cirrus 5000 HD-OCT Angioplex (Carl Zeiss Meditec, Dublin, CA, USA), fundus autofluorescence and fundus fluorescein angiography (Heidelberg Engineering, Germany). MD (mean deviation) and PSD (pattern standard deviation) parameters of 10-2 and 30-2 visual field (VF) testing strategies with a Humphrey Field Analyzer model 750I (Carl Zeiss Meditec, Dublin, CA, USA) were obtained. The electrophysiological function was assessed with mfERG evaluation (Monpack 3, Metrovision, France) according to the International Society for Clinical Electrophysiology of Vision (ISCEV) guidelines [27]. BCVA was converted to the logarithm of the minimal angle of resolution (logMAR) equivalent.

The patients were excluded from the study, if they had 1) coexisting ocular pathology that may affect visual acuity, visual field and retinal morphology such as glaucoma, uveitis, previous vitreoretinal surgery, 2) coexisting cataract that may affect mfERG, visual field and/or ocular imaging, 3) refractive error that may affect measurements higher than +6.00D, lower than -6.00D 4) coexisting systemic diseases that may affect visual function such as diabetes, vasculitis, rheumatological diseases and chronic immunosuppressive use, 5) periocular injection of platelet-rich blood and transcorneal electrical stimulation in previous 6 months and 6) previous ocular surgery.

Electrophysiologic Testing After 30 minutes of dark adaptation and pupil dilatation with the application of one drop of tropicamide 1% (Tropamid, Bilim ˙Ilaç, Turkey), phenylephrine 2.5% (Mydfrin, Alcon), and proparacaine hydrochloride 0.5% (Alcaine, Alcon), ERG jet electrodes were placed. Multifocal electroretinographies were recorded after pupil dilatation. The stimulated retinal area was subtended in an area of 60° x 55°; 61 hexagon stimulants were used with alternating black (5 cd/m2) and white (100 cd/m2) stimulants. The concentric rings were analyzed according to International Society for Clinical Electrophysiology of Vision standards.13 The amplitude and latencies of P1, N1, and N2 components were recorded for every ring. The mean signal amplitudes (MSAs) of multifocal electroretinography (mfERG) in the macula (central 0°-2°) and the peripheral (2°-5°,5°-10°, 10°-15°, and >15°) signal amplitude changes were evaluated separately.

Spheroidal Stem Cell Preparation First passage umbilical cord-derived mesenchymal stem cell was obtained from Labcell Cellular Laboratory Center which provides GMP (good manufacturing practices) conditions.

Spheroid Production The spheroid production continued in GMP condition. First passage umbilical cord-derived mesenchymal stem cells were used in the production of spheroids. 100,000 mesenchymal stem cells were suspended with 100 μl. Serum-free medium (MSC NutriStem® XF Medium, Sartorius) containing %1 ciprofloxacin (Polipharma). Each well of the low-attachment 96 well plate was seeded with 100,000 cells in 100 μl. medium. The cells were incubated at 37 °C for 48 hours. At the end of 48 hours, all spheroids were collected with a micropipette and transferred into Ringer's lactate solution (Osel/ Biofleks) containing 1% HSA (csl behring). Spheroids were washed 3 times with Ringer's lactate solution containing 1% HAS (csl behring). 50 spheroids were produced for one patient (50 spheroids containing 5x106 cells were produced). 5 of 50 spheroids were reserved for quality control analysis. The remaining 45 spheroid membranes were embedded in the matrix.

Matrix Production and Cell Embedding Culture Matrix mixture containing 225 µl cryoprecipitate + 22.5 µl calcium (Adeka) + 2.5 µl transamine (Haver) was added to each well of the 96 well plates. When the matrix became semi-solid, 45 spheroids were embedded in the middle of the matrix and incubated at 37 °C for 45 min. The matrix, which became completely solid after 45 minutes, was removed with the help of a scalpel, transferred into Ringer's lactate solution (Osel/ Biofleks) containing 1% HAS (csl behring), and transferred to the operating room in this solution (Figure 1).

Quality Control Analysis Microbiological blood culture, fungal, endotoxin analysis and purity (ciprofloxacin <0,1 µg/ml), efficiency (adipocyte and cartilage differentiation analysis) Cell Count/Viability and flow cytometric analysis (CD34 <%2, CD45 <%4, CD90 >%80, HLA-DR <%4, CD105 >%60, CD73 >%70) were studied from the reserved spheroids for quality control analyses.

Surgical Technique Patients underwent surgery under general anesthesia. The inferotemporal quadrant was chosen as the surgical area. 6.0 silk was used as the anchoring suture near the limbus between 4 and 5 o'clock. Conjunctiva and tenon were opened as 6 mm long cut at 6 mm from limbus parallel to the limbus and the edges of the cut were advanced 3 mm posteriorly. Two 8.0 vicryl sutures were used as traction sutures at the anterior corners of the conjunctiva. The tenon was dissected over the sclera posteriorly. Then we performed a 7x7 scleral flap. Anterior margin of the scleral flap was created at 8 mm from the limbus, parallel to the limbus with 30 degrees ophthalmic knife. Two other half-thickness side cuts were made to create a U-shaped flap that has its base parallel to the lateral rectus muscle. Then starting from the infero-anterior edge, a deep scleral flap was dissected with a crescent blade. During the dissection black choroidal reflex should be observed all around the surface of the flap bed. The fibrin plug carrying spheroidal stem cells was placed over the choroid that was seen under the thin sclera. It was covered by the scleral flap and the flap was sutured to its original position from its edges with a 7.0 vicryl suture. Tenon and conjunctiva were closed separately with an 8.0 vicryl suture.

ELIGIBILITY:
Inclusion Criteria:

1) Clinical and genetic diagnosis of Retinitis Pigmentosa

Exclusion Criteria:

1. Coexisting ocular pathology that may affect visual acuity, visual field and retinal morphology such as glaucoma, uveitis, previous vitreoretinal surgery,
2. Coexisting cataract that may affect mfERG, visual field and/or ocular imaging,
3. Refractive error that may affect measurements higher than +6.00D, lower than -6.00D
4. Coexisting systemic diseases that may affect visual function such as diabetes, vasculitis, rheumatological diseases and chronic immunosuppressive use,
5. Periocular injection of platelet-rich blood and transcorneal electrical stimulation in previous 6 months and 6) previous ocular surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Change in visual acuity after stem cell implantation in Retinitis Pigmentosa | 3 years
  Pre-implantation and post-implantation BCVA was converted to the logarithm of the minimal angle of resolution (logMAR) equivalent.
Change in microperimetric evaluation after stem cell implantation in Retinitis Pigmentosa | 3 years
  MD (mean deviation) and PSD (pattern standard deviation) parameters of 10-2 and 30-2 visual field (VF) testing strategies with a Humphrey Field Analyzer model 750I (Carl Zeiss Meditec, Dublin, CA, USA) were obtained.
Change in electrophysiological testing after stem cell implantation in Retinitis Pigmentosa | 3 years
  The electrophysiological function was assessed with mfERG evaluation (Monpack 3, Metrovision, France) according to the International Society for Clinical Electrophysiology of Vision (ISCEV) guidelines.After 30 minutes of dark adaptation and pupil dilatation with the application of one drop of tropicamide 1% (Tropamid, Bilim ˙Ilaç, Turkey), phenylephrine 2.5% (Mydfrin, Alcon), and proparacaine hydrochloride 0.5% (Alcaine, Alcon), ERG jet electrodes were placed. Multifocal electroretinographies were recorded after pupil dilatation. The concentric rings were analyzed according to International Society for Clinical Electrophysiology of Vision standards. The amplitude and latencies of P1, N1, and N2 components were recorded for every ring. The mean signal amplitudes (MSAs) of multifocal electroretinography (mfERG) in the macula (central 0°-2°) and the peripheral (2°-5°,5°-10°, 10°-15°, and >15°) signal amplitude changes were evaluated separately.

CONTACTS AND LOCATIONS:
Overall Officials: Berna Özkan, Professor, Principal Investigator — Acibadem University; Ercüment Ovalı, Professor, Study Chair — Acıbadem LabCell Cellular Therapy Center
Locations (1):
- Acıbadem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No